CLINICAL TRIAL: NCT02053155
Title: Development and Implementation of a Peri Operative Smoking Cessation Program With Computer Based Patient Education.
Brief Title: Peri Operative Smoking Cessation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6/11/2013; NCT01904370 (obsolete NCT alias)
Record Dates: First submitted 2014-01-31; First posted 2014-02-03 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; perioperative complication; Smokerlyzer; smokers help line
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- computer based patient education (Experimental): The patients will complete a pre module and post module set of questions to determine whether their knowledge about peri operative smoking cessation increase smoking has changed. According to their willingness and eligibility, pharmacotherapy will be given.
  Interventions: Behavioral: Computer based patient education

INTERVENTIONS:
Behavioral: Computer based patient education

SUMMARY:
Implementation of a perioperative smoking cessation program with computer based patient education increases the rate of short term (1 month) and long term (6 month) reduces the incidence of perioperative complications in elective surgical patients.

DETAILED DESCRIPTION:
Patients will be enrolled in the quit smoking before surgery program. Before participating in the education program, the investigators will ask patients questions about their smoking habits, and patient will complete pre-education questionnaires that should take about 5 minutes. Patients will participate in a computer-based education program about quitting smoking for about 15 minutes. It will explain the importance of quitting smoking before their surgery, how to quit and coping with quitting. If they are not familiar with using a computer, we will provide an assistant for them to complete the education program. After completing the education program, they will complete a post-education questionnaire. patients will also receive an information pamphlet.

All participants will receive the computer-based education program, brief counselling, pamphlet, Smokers' Helpline referral, and telephone follow-up.

Altogether you will be spending about 30 minutes to complete the assessment, education program and counselling.

patients will be asked for their permission to inform their family physician about their participation in this study. Their smoking status, date of surgery, quit date, and recommended medication (when appropriate) will be faxed to your family physician to assist them quitting process. If they are willing to accept the assistance from Smokers' Helpline, their name and phone number will be faxed to the Smokers' Helpline, and someone from Smokers' Helpline will call you in the next 48 hours to follow-up.

The investigators will monitor patient's smoking behavior by measuring expired carbon monoxide, a gas in the air they breathe out, during their pre-surgery visit and on the day of surgery. We also will measure urine cotinine (a by-product of nicotine) by taking urine samples and check their smoking status by asking questions about their smoking habits on the day of surgery, 1 month, 3 months and 6 months after their surgery. During the telephone interview follow-up, we will remind them to do the urine cotinine and mail it to us. (Prepaid mail with urine cotinine strip will be provided at the time of the 2nd visit on the day of surgery.) Each follow-up phone call will take about 6 -10 minutes.

A one-month,3 month and 6 month follow up will be done by the research coordinator to assess the smoking status. Brief counseling (< 5 mins) will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients> 18 years of age
* self reported smokers ( daily or non daily smokers)
* Scheduled for elective surgical procedures

Exclusion Criteria:

* patients who cannot read and understand English
* Have any form of cognitive impairment
* Do not have a telephone
* Drug or alcohol abuser dependence within the past year
* Patients whop are already on pharmacotherapy for smoking cessation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Quit rate | 6 month
  we will do urine cotinine analysis to confirm the abstinence

SECONDARY OUTCOMES:
Surgical outcome | 1 month
  we will do a chart review to find out the intraoperative and post operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wong, FRCPC, Principal Investigator — Associate professor, dewpartment of anesthesia. Toronto Western Hospital, University Health Network, University of Toronto, Toronto, Ontario
Locations (3):
- Canada (3):
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Womens College Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Wong J, Raveendran R, Chuang J, Friedman Z, Singh M, Patras J, Wong DT, Chung F. Utilizing Patient E-learning in an Intervention Study on Preoperative Smoking Cessation. Anesth Analg. 2018 May;126(5):1646-1653. doi: 10.1213/ANE.0000000000002885. PMID 29517567